CLINICAL TRIAL: NCT03491449
Title: Intensive Treatment of Blood Pressure in Acute Ischemic Stroke. Study TICA 2
Acronym: TICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manuel Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Manuel Rodríguez, Principal Investigator, Hospital Clinico Universitario de Santiago
Organization: Hospital Clinico Universitario de Santiago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRY-IIA-2015-01
Record Dates: First submitted 2018-03-06; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Brain Ischemia
Keywords: Brain ischemia; Cerebral ischemia
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Intervention Model Description: National, multicenter, open, two-parallel groups, randomized 1: 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: pressure ≥140 and ≤160mmHg (Experimental): Intensive management of blood pressure, maintaining a systolic blood pressure ≥ 140 and ≤ 160 mm Hg for 72 hours.
  Interventions: Procedure: Group A
- Group B: Keep systolic pressure <185mmHg (Active Comparator): Intensive management of blood pressure, maintaining systolic blood pressure <185 mm Hg for 72 hours.
  Interventions: Procedure: Group B

INTERVENTIONS:
Procedure: Group A — Maintaining a systolic blood pressure ≥ 140 and ≤ 160mm Hg for 72 hours.
  Arms: Group A: pressure ≥140 and ≤160mmHg
Procedure: Group B — Maintaining a systolic blood pressure <185mm Hg for 72 hours.
  Arms: Group B: Keep systolic pressure <185mmHg

SUMMARY:
Demonstrate that maintenance of systolic blood pressure between 140 and 160 mm Hg during the acute phase of ischemic stroke is more effective than management according to the International Guideline (treat when systolic blood pressure exceeds 185 mm Hg)

DETAILED DESCRIPTION:
Control of blood pressure figures remains one of the most important risk factors in primary and secondary prevention in patients with stroke. The current strategy for the hypertensive treatment of patients during the acute phase of ischemic stroke within the first 72 hours remains a highly debated and unclear issue, with no consensus on the range or appropriate blood pressure ranges to be handled (13).

Team study working hypothesis focuses on the study of blood pressure (for 72 hours), through its intensive control (recording and adjustment every four hours), in the acute phase of ischemic stroke. Specifically, it is based on the monitoring and maintenance of systolic blood pressure between 140 and 160 mm Hg in patients with acute ischemic stroke; And this can lead to a better functional prognosis, measured at 90 days, compared with the functional prognosis of patients treated according to the recommendations of the current Clinical Guidelines, which propose to act on systolic blood pressure only when it exceeds 185 mm Hg (13,22).

Although the intense decrease in blood pressure during the acute phase of stroke has the potential risk of decreasing cerebral perfusion in the area of ischemic penumbra, in recent observational studies (19), a worse functional prognosis has not been found in those patients With systolic blood pressure above 140 mm Hg.

There is no previous evidence from other intervention studies related to blood pressure control and a benefit to patients with acute ischemic stroke. Comparison using a randomized clinical trial of a group of patients with blood pressure control following current guidelines with a group of patients with systolic blood pressure between 140 and 160 mm Hg may allow a simple, rapidly applicable therapeutic alternative to Clinical practice, low cost and extrapolable to a wider population, such as patients with stroke of any etiology.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and up to and 85 years (both included).
* Clinical and neuroimaging diagnosis (CT or MRI) of ischemic stroke.
* Possibility of initiating antihypertensive treatment within 12 hours after the onset of symptoms (in the case of stroke, the start time is considered the time in that the patient has been seen asymptomatic for the last time).
* Participant with systolic blood pressure greater than or equal to 140 mm Hg and less than or equal to 220 mm Hg at the time of inclusion.
* Participant or legal representative able to understand the study requirements and sign Informed consent.

Exclusion Criteria:

* Uncontrollable hypertension (SBP greater than 220 mm Hg) or any condition requiring urgent antihypertensive treatment.
* Have suffered a stroke in the previous 90 days in the same territory as the current stroke.
* Had a myocardial infarction in the previous 90 days.
* Suspected aortic dissection or hypertensive encephalopathy.
* Presence of intracerebral or subarachnoid hemorrhage in basal neuroimaging (Computed tomography or magnetic resonance imaging).
* Recanalization is possible or intraarterial recanalization techniques have been performed due to the current stroke.
* Known critical carotid occlusion or stenosis.
* To be a candidate for carotid revascularization in the next three months.
* Previous alterations that, in the opinion of the investigator, may interfere in the interpretation of the neurological scales.
* Coma or low level of consciousness (defined as a score ≥ 2 in section 1.a of NIHSS), dementia or mental disability that, in the opinion of the investigator, patient is unable to participate in the study.
* Convulsive seizures at any time from the onset of symptoms to the initial evaluation.
* Neurological or non-neurological comorbidities that, in the opinion of the investigator, may lead, regardless of the current stroke, to a deterioration in the patient's neurologic status during the study period, or may hinder the evaluation of the neurological state caused only by stroke (i.e., metabolic encephalopathies, hemiplegic migraine, multiple sclerosis, central nervous system tumor, epilepsy, monocular blindness).
* Patient is likely to undergo a procedure involving extracorporeal circulation during the study period.
* Any condition that, in the opinion of the investigator, may compromise the patient's ability to complete the study (i.e., concomitant diseases that may threaten the patient's life, such as neoplasms or terminal failure of an organ).
* Patient's previous disability, determined by a score in modified Rankin scale > 1.
* Women of childbearing age with positive pregnancy test or breastfeeding at the time of inclusion.
* Women of childbearing potential (menopause less than 2 years old or not surgically sterilized) who are not going to take effective and adequate measures to avoid conception during the study period. Control measures include hormonal contraceptives, barrier methods such as diaphragm or intrauterine devices and / or spermicidal preservatives.
* Current dependence on substances of abuse such as alcohol, sympathomimetic amines, cannabis, cocaine, hallucinogens, opioids, phencyciclin, sedatives or hypnotics.
* Life expectancy is less than the expected duration of the clinical trial or any situation that, at the discretion of the investigator, may make participation in the clinical trial dangerous (eg drug use, alcohol addiction, etc.).
* Have received a drug or product under or participate in a clinical trial within 30 days prior to the date of inclusion in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-02-13 (Estimated); Study Completion 2020-02-13 (Estimated)

PRIMARY OUTCOMES:
Study of functional prognosis in patients with acute ischemic stroke using modified Rankin | 90 days
  Study of functional prognosis in patients with acute ischemic stroke using modified Rankin scale measured at 90 ± 15 days will compared between the two branches.Rankin Scale: It is a scale that evaluates the patient's functional situation. The full name is "modified Rankin Scale", and the abbreviated name is "mRS". The range of the scale is from 0 to 6, where 0 is the best score (the patient is asymptomatic) and 6 is the worst score (mortality). Up to 2 the patient is considered independent, and from 3 the patient needs help for the activities of daily life.

SECONDARY OUTCOMES:
Early Neurological Impairment (ENI) | 72 hours
  Increased at 4 or more points on the NIHSS scale in any determination during the first 72 hours compared to baseline score. NIHSS Scale: It is a scale that evaluates the neurological situation of the patient. The full name is "National Institute of Health Stroke Scale." The lowest score is 0, and the upper limit is 40. The lower score, the patient has fewer symptoms, and the higher score, the patient is more serious. It is considered that up to 8 points the patient has a mild stroke, between 8-15 a moderate stroke and more than 16 points a severe stroke.
Volume of the infarct in neuroimaging | 4th day
  Volume of the infarct in neuroimaging (CT or MRI) performed between the 4th and 7th day after the stroke. The volume in mL, using the formula a x b x c x 0.5, where "a" and "b" are the largest diameters perpendicular in centimeters and "c" the number of 1 cm cuts in which the infarct is seen.
Mortality | 90 days
  Any patient who dies from inclusion (signature of informed consent) until the final study visit (90 ± 15 days).
Measuring the adverse events | 90 days
  Measuring the adverse events occurring throughout the study.
Volume of the infarct using NIHSS | 7th day
  Increased at 4 or more points on the NIHSS scale in any determination during the first 72 hours compared to baseline score. NIHSS Scale: It is a scale that evaluates the neurological situation of the patient. The full name is "National Institute of Health Stroke Scale." The lowest score is 0, and the upper limit is 40. The lower score, the patient has fewer symptoms, and the higher score, the patient is more serious. It is considered that up to 8 points the patient has a mild stroke, between 8-15 a moderate stroke and more than 16 points a severe stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodríguez, MD, Principal Investigator — Hospital Universitario de Santiago
Locations (3):
- Spain (3):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario A Coruña, A Coruña

IPD SHARING:
Plan to Share IPD: No